CLINICAL TRIAL: NCT01492712
Title: Validation Study of Covariates Model (VaSCoM) for Propofol
Acronym: VaSCoM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Golden Jubilee National Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: VaSCoM005; 2009-017900-10 (EudraCT Number)
Record Dates: First submitted 2011-12-08; First posted 2011-12-15 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Target Controlled Infusion of Propofol
Keywords: Propofol; Pharmacokinetics; Pharmacodynamics; Infusion Pumps
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-high-low blood target concentration (Experimental): Patients in the low-high-low group will receive an infusion of propofol with an initial blood target concentration of 2 mcg/ml. After 15 minutes the target will be increased to 5 mcg/ml and after a further 15 minutes the target will be reduced back to 2 mcg/ml for a further 15 to 30 minutes.
  Interventions: Drug: Propofol
- High-low-high target blood concentration (Experimental): Patients in the high-low-high group will receive an infusion of propofol with an initial blood target concentration of 5 mcg/ml. After 15 minutes the target will be reduced to 2 mcg/ml and after a further 15 minutes the target will be increased back to 5 mcg/ml for a further 15 to 30 minutes.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Patients in the low-high-low group will receive an infusion of propofol with an initial blood target concentration of 2 mcg/ml. After 15 minutes the target will be increased to 5 mcg/ml and after a further 15 minutes the target will be reduced back to 2 mcg/ml for a further 15 to 30 minutes.
  Arms: Low-high-low blood target concentration
Drug: Propofol — Patients in the high-low-high group will receive an infusion of propofol with an initial blood target concentration of 5 mcg/ml. After 15 minutes the target will be reduced to 2 mcg/ml and after a further 15 minutes the target will be increased back to 5 mcg/ml for a further 15 to 30 minutes.
  Arms: High-low-high target blood concentration

SUMMARY:
Anaesthesia for surgical procedures can be provided using a continuous infusion of intravenous drug. The most commonly used drug for this technique is propofol. Infusion devices programmed with pharmacokinetic models can be used to infuse propofol to achieve a target blood concentration. These pharmacokinetic models predict the rate of distribution of propofol within the body and also the rate at which it is cleared. In practice, the anaesthetist enters patient details such as age, sex and weight as well as a target blood concentration of propofol. The infusion device then infuses propofol at the appropriate rate to achieve this concentration.

White and colleagues recently published the Covariates Model for propofol. It is anticipated that this model will have reduced bias and inaccuracy compared to the models in current clinical use. The VaSCoM study has three objectives:

1. Prospective validation of the Covariates Model
2. Modelling of the effect site concentration of propofol
3. Comparison of propofol concentration in venous and arterial blood samples

To achieve the above objectives, patients over 18 years of age and undergoing elective non-cardiac surgery will be recruited to the study. Anaesthesia will be delivered using a target controlled infusion device programmed with the Covariates Model for propofol. The target blood concentrations will be set according to a pre-determined schedule and all measurements will be made prior to the start of surgery.

Prospective validation of the Covariates Model will be done by comparing blood concentration of propofol predicted by the model to those actually measured. These results will then be compared to the predictions made using the models in current clinical practice.

Modelling of the effect site means predicting the concentration of propofol in the brain for a given blood concentration. This will involve using depth of anaesthesia monitors (such as bispectral index) as surrogate markers of brain concentration and comparing this to the predicted and measured blood concentrations of propofol.

Finally, important information on the distribution and clearance of propofol can be gained through the comparison of venous and arterial blood samples. In this study, simultaneous sampling of venous and arterial blood will facilitate this comparison.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* ASA I/II
* Elective non-cardiac surgery expected to last longer than 30 minutes

Exclusion Criteria:

* Patient refusal or unable to consent
* Premedication, sedative or anaesthetic in the previous 12 hours
* Pre-operative GCS less than 15
* ASA III/IV
* Allergy to constituents of propofol
* Excess alcohol intake
* Drug abuse
* Mental retardation
* Difficult airway
* BMI over 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Performance error of predicted blood propofol concentration (venous blood samples) | 1.5, 5, 16.5, 20, 31.5, 35, 45-60 minutes post infusion start time
  Performance error is calculated as:
  ((Measured blood concentration - Predicted blood concentration)/ Predicted blood concentration) x 100
  The median performance error and the absolute performance error can then be calculated as measures of bias and inaccuracy respectively.

SECONDARY OUTCOMES:
Depth of anaesthesia | 0 to 45-60 minutes post infusion start time
  Depth of anaesthesia (as measured by bispectral index and index of consciousness) will be used as a surrogate marker of propofol effect site concentration. By using complex statistical analysis to compare depth of anaesthesia to measured and predicted blood concentrations, we aim to determine the Keo. This is the rate constant for elimination of propofol from the effect site compartment and will be incorporated to the Covariates Model to predict brain concentration for a given blood concentration of propofol.
Comparison of performance errors calculated from venous blood samples to performance errors calculated from arterial blood samples | 1.5, 5, 16.5, 20, 31.5, 35, 45-60 minutes post infusion start time
  Performance error is calculated as:
  ((Measured blood concentration - Predicted blood concentration)/ Predicted blood concentration) x 100

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schraag, Principal Investigator — Golden Jubilee National Hospital
Locations (1):
- Golden Jubilee National Hospital, Clydebank, United Kingdom

REFERENCES:
- [Derived] Hawthorne C, Shaw M, Campbell R, Sutcliffe N, McKelvie S, Schraag S. Clinical Validation of the Covariates Pharmacokinetic Model for Propofol in an Adult Population. Drugs R D. 2022 Dec;22(4):289-300. doi: 10.1007/s40268-022-00404-4. Epub 2022 Oct 7. PMID 36207643